CLINICAL TRIAL: NCT02738515
Title: Clinical Efficacy of Subgingivally Delivered 0.75% Boric Acid Gel as an Adjunct to Mechanotherapy in Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Boric Acid in Degree 2 Furcation Defect
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor & Head, Department of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014ZM
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Periodontitis With Mandibular Degree 2 Furcation Defects
MeSH Terms: interventions — boric acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 (Active Comparator): Scaling and Root Planing (SRP) with 0.75% BORIC ACID GEL for treating furcation defect
  Interventions: Drug: 0.75 % Boric Acid
- Group 2 (Placebo Comparator): Scaling and Root Planing (SRP) with PLACEBO GEL for treating furcation defect.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 0.75 % Boric Acid — After Scaling and Root Planing placement of 0.75% Boric Acid gel in Mandibular degree 2 Furcation defect.
  Arms: Group 1
Drug: placebo — After Scaling and Root Planing placement of Placebo gel in Mandibular degree 2 Furcation defect.
  Arms: Group 2

SUMMARY:
The purpose of this double-masked, randomized, controlled clinical trial was to evaluate the effects of subgingival delivery of boric acid gel as an adjunct to scaling and root planing (SRP) on clinical and radiographic parameters and compare this method with SRP plus placebo gel alone in patients with chronic periodontitis (CP).

DETAILED DESCRIPTION:
Background: The purpose of this double-masked, randomized, controlled clinical trial was to evaluate the effects of subgingival delivery of boric acid gel as an adjunct to scaling and root planing (SRP) on clinical and radiographic parameters and compare this method with SRP plus placebo gel alone in patients with chronic periodontitis (CP).

Methods:FORTY EIGHT systemically healthy patients with CP are included in this study. They were divided into two groups: 1) SRP + 0.75% Boric acid gel (BA group); 2) SRP + Placebo gel (Placebo group). At baseline, 3 month, and 6 months after treatment, clinical measurements, including plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), clinical attachment level (CAL) and radiographic parameters intrabony defect depth (IBD), percentage change in radiographic defect depth reduction (DDR%) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of buccal Class II furcation defects in endodontically vital, asymptomatic mandibular first and second molars with a radiolucency in the furcation area on an intraoral periapical radiograph with probing depth (PD) ≥ 5mm and horizontal ≥ PD 3mm after phase I therapy i.e, scaling and root planing (SRP)
* No history of antibiotic or periodontal therapy in the preceding 6 months

Exclusion Criteria:

* Systemic conditions known to affect the periodontal status
* Medications known to affect the outcomes of periodontal therapy
* Hematological disorders and insufficient platelet count (<200,000/mm3)
* Pregnancy/lactation
* Smoking and tobacco use in any form
* Immunocompromised individuals
* Those having unacceptable oral hygiene (plaque index [PI] >1.5)
* Teeth with furcation involvement, non-vital teeth, and carious teeth indicated for restorations and mobility of at least grade II
* Aggressive periodontitis

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Radiographic bone fill | Baseline to 6 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth | 3 and 6 months
  measured in mm
Relative vertical attachment leve | 3 and 6 months
  measured in mm
Relative horizontal attachment level | 3 and 6 months
  measured in mm
modified sulcus bleeding index | 3 and 6 months
  0-3 scale
plaque index | 3 and 6 months
  0-3 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India